CLINICAL TRIAL: NCT01790243
Title: A Prospective, Multicenter, Registry of the Lutonix Drug Coated Balloon for Treatment of Femoropopliteal Arteries (LEVANT 2 Safety Registry)
Brief Title: LEVANT 2 Safety Registry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL0006-01
Record Dates: First submitted 2013-02-08; First posted 2013-02-13 (Estimated); Results first posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-05

CONDITIONS: Peripheral Artery Disease; Femoropopliteal Artery Occlusion; Femoropopliteal Stenosis
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lutonix Drug Coated Balloon (Experimental): Formerly called the Moxy Drug Coated Balloon, the Lutonix Drug Coated Balloon (Lutonix DCB) is a paclitaxel coated balloon catheter
  Interventions: Device: Lutonix Drug Coated Balloon
- Standard Uncoated Angioplasty Balloon (Active Comparator): PTA Catheter
  Interventions: Device: Standard PTA Balloon

INTERVENTIONS:
Device: Lutonix Drug Coated Balloon — Use of the Lutonix Drug Coated Balloon (DCB) for the treatment of stenosis or occlusion of the femoropopliteal arteries.
  Arms: Lutonix Drug Coated Balloon
Device: Standard PTA Balloon — Use of Standard PTA Balloon in the treatment of stenosis or occlusion of the femoropopliteal arteries.
  Arms: Standard Uncoated Angioplasty Balloon

SUMMARY:
The primary objective of the LEVANT 2 Extended Follow-up Post-Approval Study (PAS 1) is to evaluate the long-term performance of the Lutonix Drug Coated Balloon (DCB) versus Percutaneous Transluminal Balloon Angioplasty (PTA) in the treatment of stenosis or occlusion of the femoropopliteal arteries.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Male or non-pregnant female ≥18 years of age;
2. Rutherford Clinical Category 2-4;
3. Patient is willing to provide informed consent, is geographically stable and comply with the required follow up visits, testing schedule and medication regimen;

   Angiographic Lesion Inclusion Criteria:
4. Length ≤15 cm;
5. Up to two focal lesions or segments within the designated 15 cm length of vessel may be treated (e.g. two discrete segments, separated by several cm, but both falling within a composite length of <15 cm);
6. ≥70% stenosis by visual estimate;
7. Lesion location starts ≥1 cm below the common femoral bifurcation and terminates distally ≤2 cm below the tibial plateau AND ≥1 cm above the origin of the TP trunk;
8. De novo lesion(s) or non-stented restenotic lesion(s) >90 days from prior angioplasty procedure;
9. Lesion is located at least 3 cm from any stent, if target vessel was previously stented;
10. Target vessel diameter between ≥4 and ≤6 mm and able to be treated with available device size matrix;
11. Successful, uncomplicated (without use of a crossing device) antegrade wire crossing of lesion;
12. A patent inflow artery free from significant lesion (≥50% stenosis) as confirmed by angiography (treatment of target lesion acceptable after successful treatment of inflow artery lesions); NOTE: Successful inflow artery treatment is defined as attainment of residual diameter stenosis ≤30% without death or major vascular complication.
13. At least one patent native outflow artery to the ankle, free from significant (≥50%) stenosis as confirmed by angiography that has not previously been revascularized (treatment of outflow disease is NOT permitted during the index procedure);
14. Contralateral limb lesion(s) cannot be treated within 2 weeks before and/or planned 30 days after the protocol treatment in order to avoid confounding complications;
15. No other prior vascular interventions within 2 weeks before and/or planned 30 days after the protocol treatment.

Exclusion Criteria:

Patients will be excluded if ANY of the following conditions apply:

1. Pregnant or planning on becoming pregnant or men intending to father children;
2. Life expectancy of <5 years;
3. Patient is currently participating in an investigational drug or other device study or previously enrolled in this study; NOTE: Enrollment in another clinical trial during the follow up period is not allowed.
4. History of hemorrhagic stroke within 3 months;
5. Previous or planned surgical or interventional procedure within 2 weeks before or within 30 days after the index procedure;
6. History of MI, thrombolysis or angina within 2 weeks of enrollment;
7. Rutherford Class 0, 1, 5 or 6;
8. Renal failure or chronic kidney disease with MDRD GFR ≤30 ml/min per 1.73 m2 (or serum creatinine ≥2.5 mg/L within 30 days of index procedure or treated with dialysis);
9. Prior vascular surgery of the index limb, with the exception of remote common femoral patch angioplasty separated by at least 2 cm from the target lesion;
10. Inability to take required study medications or allergy to contrast that cannot be adequately managed with pre- and post-procedure medication;
11. Anticipated use of IIb/IIIa inhibitor prior to randomization;
12. Ipsilateral retrograde access;
13. Composite lesion length is >15 cm or there is no normal proximal arterial segment in which duplex flow velocity can be measured;
14. Significant inflow disease. Successful treatment of inflow disease allowed prior to target lesion treatment;
15. Known inadequate distal outflow (>50 % stenosis of distal popliteal and/or all three tibial vessels), or planned future treatment of vascular disease distal to the target lesion;
16. Sudden symptom onset, acute vessel occlusion, or acute or sub-acute thrombus in target vessel;
17. Severe calcification that renders the lesion un-dilatable;
18. Use of adjunctive treatment modalities (i.e. laser, atherectomy, cryoplasty, scoring/cutting balloon, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1189 (Actual)
Dates: Start 2011-07-20 (Actual); Primary Completion 2015-11-27 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Rosenfield, MD, Principal Investigator — Massachusetts General Hospital
Locations (8):
- United States (8):
  - Mission Cardiovascular Research Institute, Fremont, California
  - Metro Health Hospital, Wyoming, Michigan
  - Jackson Heart Clinic/St. Dominic's Hospital, Jackson, Mississippi
  - Mercy Hospital, Springfield, Missouri
  - Holy Name Medical Center, Teaneck, New Jersey
  - New York Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - TriHealth Heart Institute, Cincinnati, Ohio
  - Mission Research Institute, New Braunfels, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lutonix Drug Coated Balloon | Standard Uncoated Angioplasty Balloon
Started | 1029 | 160
Completed | 739 | 117
Not Completed | 290 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lutonix Drug Coated Balloon | Standard Uncoated Angioplasty Balloon | Total
Number analyzed (Participants) | 1029 | 160 | 1189
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.4 (9.7) | 69.0 (9) | 68.48 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 383 | 53 | 436
  Male | 646 | 107 | 753
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 14 | 53
  Not Hispanic or Latino | 988 | 146 | 1134
  Unknown or Not Reported | 2 | 0 | 2
Baseline Rutherford Classification [Count of Participants; unit: Participants] — Measure Description: Rutherford Classification is on an ascending scale from 0 to 6. Lower classifications on the scale indicate more favorable outcomes.
  0- Asymptomatic
  1. Mild claudication
  2. Moderate claudication
  3. Severe claudication
  4. Rest pain
  5. Ischemic ulceration not exceeding ulcer of the digits of the foot
  6. Severe ischemic ulcers or frank gangrene
  Participants
    Rutherford 0 | 0 | 0 | 0
    Rutherford 1 | 0 | 0 | 0
    Rutherford 2 | 354 | 55 | 409
    Rutherford 3 | 606 | 92 | 698
    Rutherford 4 | 69 | 13 | 82
    Rutherford 5 | 0 | 0 | 0
    Rutherford 6 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Unanticipated Device- or Drug-Related Serious Adverse Events at 60 Months Post Index Procedure.
Time Frame: From index procedure to 60 months Post Index Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix Drug Coated Balloon | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 1029 | 160
Participants | 0 | 0

2. Secondary Outcome: Number of Subjects With Freedom From Death, Index-Limb Amputation, and Target Vessel Revascularization (TVR) at 30 Days Post Index Procedure
Description: Number of subjects with Freedom from all-cause death, index limb amputation above the ankle and Target Vessel Revascularization (TVR) (VIVA Safety Endpoint)
Time Frame: 30 days post index procedure
Population: The number of participants (n) varies from the total number of participants (N) in the study as n depends on the number of participants for which data was available at the given time-point analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix Drug Coated Balloon | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 1009 | 156
Participants | 1002 | 155

3. Secondary Outcome: Number of Participants With All-Cause Perioperative (<30 Day) Death, Index Limb Amputation, Index Limb Re-intervention, and Index Limb Related Death at 1,6, 12, 24, 36, 48, and 60 Months Post Index Procedure
Time Frame: 1, 6, 12, 24, 36, 48, and 60 months post index procedure (PPI)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lutonix Drug Coated Balloon | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 1010 | 156
participants
  Death : 1 month post index procedure: number analyzed (Participants) | 1009 | 156
  Death : 1 month post index procedure | 1 | 0
  Death : 6 months post index procedure: number analyzed (Participants) | 990 | 154
  Death : 6 months post index procedure | 8 | 2
  Death : 12 months post index procedure: number analyzed (Participants) | 967 | 148
  Death : 12 months post index procedure | 18 | 4
  Death : 24 months post index procedure: number analyzed (Participants) | 927 | 141
  Death : 24 months post index procedure | 46 | 8
  Death : 36 months post index procedure: number analyzed (Participants) | 912 | 139
  Death : 36 months post index procedure | 82 | 10
  Death : 48 months post index procedure: number analyzed (Participants) | 901 | 137
  Death : 48 months post index procedure | 121 | 14
  Death : 60 months post index procedure: number analyzed (Participants) | 879 | 133
  Death : 60 months post index procedure | 147 | 17
  Major Amputation : 1 month post index procedure: number analyzed (Participants) | 1008 | 156
  Major Amputation : 1 month post index procedure | 0 | 0
  Major Amputation : 6 months post index procedure: number analyzed (Participants) | 982 | 153
  Major Amputation : 6 months post index procedure | 1 | 0
  Major Amputation : 12 months post index procedure: number analyzed (Participants) | 955 | 144
  Major Amputation : 12 months post index procedure | 1 | 0
  Major Amputation : 24 months post index procedure: number analyzed (Participants) | 890 | 134
  Major Amputation : 24 months post index procedure | 2 | 0
  Major Amputation : 36 months post index procedure: number analyzed (Participants) | 843 | 131
  Major Amputation : 36 months post index procedure | 3 | 0
  Major Amputation : 48 months post index procedure: number analyzed (Participants) | 791 | 124
  Major Amputation : 48 months post index procedure | 6 | 1
  Major Amputation : 60 months post index procedure: number analyzed (Participants) | 740 | 116
  Major Amputation : 60 months post index procedure | 8 | 1
  Minor Amputation : 1 month post index procedure: number analyzed (Participants) | 1008 | 156
  Minor Amputation : 1 month post index procedure | 1 | 0
  Minor Amputation : 6 months post index procedure: number analyzed (Participants) | 981 | 153
  Minor Amputation : 6 months post index procedure | 1 | 0
  Minor Amputation : 12 months post index procedure: number analyzed (Participants) | 954 | 144
  Minor Amputation : 12 months post index procedure | 1 | 0
  Minor Amputation : 24 months post index procedure: number analyzed (Participants) | 888 | 134
  Minor Amputation : 24 months post index procedure | 3 | 0
  Minor Amputation : 36 months post index procedure: number analyzed (Participants) | 841 | 131
  Minor Amputation : 36 months post index procedure | 5 | 0
  Minor Amputation : 48 months post index procedure: number analyzed (Participants) | 790 | 124
  Minor Amputation : 48 months post index procedure | 9 | 0
  Minor Amputation : 60 months post index procedure: number analyzed (Participants) | 737 | 116
  Minor Amputation : 60 months post index procedure | 9 | 0
  Amputation Free Survival : 1 month PPI: number analyzed (Participants) | 1009 | 156
  Amputation Free Survival : 1 month PPI | 1008 | 156
  Amputation Free Survival : 6 months: number analyzed (Participants) | 989 | 154
  Amputation Free Survival : 6 months | 981 | 152
  Amputation Free Survival : 12 months PPI: number analyzed (Participants) | 967 | 148
  Amputation Free Survival : 12 months PPI | 949 | 144
  Amputation Free Survival : 24 months PPI: number analyzed (Participants) | 928 | 141
  Amputation Free Survival : 24 months PPI | 881 | 133
  Amputation Free Survival : 36 months PPI: number analyzed (Participants) | 913 | 139
  Amputation Free Survival : 36 months PPI | 830 | 129
  Amputation Free Survival : 48 months PPI: number analyzed (Participants) | 901 | 137
  Amputation Free Survival : 48 months PPI | 776 | 122
  Amputation Free Survival : 60 months PPI: number analyzed (Participants) | 881 | 133
  Amputation Free Survival : 60 months PPI | 729 | 115
  Target Vessel Revascularization : 1 month PPI: number analyzed (Participants) | 1008 | 156
  Target Vessel Revascularization : 1 month PPI | 6 | 1
  Target Vessel Revascularization : 6 months PPI: number analyzed (Participants) | 981 | 153
  Target Vessel Revascularization : 6 months PPI | 48 | 12
  Target Vessel Revascularization : 12 months PPI: number analyzed (Participants) | 955 | 146
  Target Vessel Revascularization : 12 months PPI | 125 | 26
  Target Vessel Revascularization : 24 months PPI: number analyzed (Participants) | 898 | 138
  Target Vessel Revascularization : 24 months PPI | 207 | 39
  Target Vessel Revascularization : 36 months PPI: number analyzed (Participants) | 857 | 135
  Target Vessel Revascularization : 36 months PPI | 240 | 43
  Target Vessel Revascularization : 48 months PPI: number analyzed (Participants) | 820 | 130
  Target Vessel Revascularization : 48 months PPI | 268 | 53
  Target Vessel Revascularization : 60 months PPI: number analyzed (Participants) | 780 | 126
  Target Vessel Revascularization : 60 months PPI | 283 | 54
  Reintervention for thrombosis : 1 month: number analyzed (Participants) | 1008 | 156
  Reintervention for thrombosis : 1 month | 2 | 0
  Reintervention for thrombosis : 6 months: number analyzed (Participants) | 981 | 153
  Reintervention for thrombosis : 6 months | 2 | 1
  Reintervention for thrombosis : 12 months: number analyzed (Participants) | 954 | 144
  Reintervention for thrombosis : 12 months | 3 | 1
  Reintervention for thrombosis : 24 months: number analyzed (Participants) | 888 | 134
  Reintervention for thrombosis : 24 months | 5 | 1
  Reintervention for thrombosis: 36 months: number analyzed (Participants) | 842 | 131
  Reintervention for thrombosis: 36 months | 7 | 1
  Reintervention for thrombosis : 48 months: number analyzed (Participants) | 789 | 124
  Reintervention for thrombosis : 48 months | 7 | 1
  Reintervention for thrombosis: 60 months: number analyzed (Participants) | 738 | 116
  Reintervention for thrombosis: 60 months | 8 | 1
  Cardiovascular Hospitalization : 1 month PPI: number analyzed (Participants) | 1009 | 156
  Cardiovascular Hospitalization : 1 month PPI | 6 | 0
  Cardiovascular Hospitalization : 6 months PPI: number analyzed (Participants) | 983 | 153
  Cardiovascular Hospitalization : 6 months PPI | 53 | 3
  Cardiovascular Hospitalization : 12 months PPI: number analyzed (Participants) | 957 | 144
  Cardiovascular Hospitalization : 12 months PPI | 88 | 10
  Cardiovascular Hospitalization : 24 months PPI: number analyzed (Participants) | 900 | 135
  Cardiovascular Hospitalization : 24 months PPI | 112 | 21
  Cardiovascular Hospitalization : 36 months PPI: number analyzed (Participants) | 858 | 132
  Cardiovascular Hospitalization : 36 months PPI | 115 | 23
  Cardiovascular Hospitalization : 48 months PPI: number analyzed (Participants) | 812 | 126
  Cardiovascular Hospitalization : 48 months PPI | 115 | 23
  Cardiovascular Hospitalization : 60 months PPI: number analyzed (Participants) | 768 | 119
  Cardiovascular Hospitalization : 60 months PPI | 115 | 23
  Major Vascular Complications : 1 month PPI | 27 | 2
  Major Vascular Complications : 6 months PPI: number analyzed (Participants) | 985 | 153
  Major Vascular Complications : 6 months PPI | 39 | 4
  Major Vascular Complications : 12 months PPI: number analyzed (Participants) | 958 | 145
  Major Vascular Complications : 12 months PPI | 51 | 71
  Major Vascular Complications : 24 months PPI: number analyzed (Participants) | 902 | 135
  Major Vascular Complications : 24 months PPI | 79 | 10
  Major Vascular Complications : 36 months PPI: number analyzed (Participants) | 861 | 132
  Major Vascular Complications : 36 months PPI | 87 | 13
  Major Vascular Complications : 48 months PPI: number analyzed (Participants) | 821 | 126
  Major Vascular Complications : 48 months PPI | 92 | 13
  Major Vascular Complications : 60 months PPI: number analyzed (Participants) | 776 | 119
  Major Vascular Complications : 60 months PPI | 93 | 13

4. Secondary Outcome: Percentage of Participants With Primary Patency of the Target Lesion at 6, 12, and 24 Months Post Index Procedure
Description: Primary Patency is defined as the absence of target lesion restenosis (defined by DUS peak systolic velocity ratio (PSVR) ≥2.5) and freedom from target lesion revascularization (TLR).
Time Frame: 6, 12, and 24 months post index procedure
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix Drug Coated Balloon | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 916 | 142
Percentage of Participants
  6 months post index procedure | 81.4 [78.9 to 84.0] | 64.8 [56.9 to 72.6]
  12 months post index procedure: number analyzed (Participants) | 897 | 137
  12 months post index procedure | 66.3 [63.2 to 69.4] | 54.0 [45.7 to 62.4]
  24 months post index procedure: number analyzed (Participants) | 841 | 127
  24 months post index procedure | 54.5 [51.1 to 57.8] | 47.2 [38.6 to 55.9]

5. Secondary Outcome: Number of Acute Device Success at Time of Index Procedure
Description: Device Success was defined as the achievement of successful delivery and deployment of the study device(s) as intended at the intended target lesion, without balloon rupture or inflation/deflation abnormalities and a successful withdrawal of the study system.
Time Frame: At time of index procedure
Measure: Count of Units; unit: Devices
Units Other Than Participants: Devices
Arm/Group | Lutonix Drug Coated Balloon | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 1029 | 160
Number analyzed (Devices) | 1404 | 180
Devices | 1402 | 180

6. Secondary Outcome: Number of Participants With Technical and Procedural Success
Description: Technical Success is defined as successful access and deployment of the device and visual estimate of ≤30% diameter residual stenosis during the index procedure without deployment of a bailout stent.
  Procedural Success is defined as attainment of ≤30% residual stenosis in the treatment area by independent core lab analysis without serious adverse events during the index procedure.
Time Frame: At time of index procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix Drug Coated Balloon | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 1016 | 159
Participants
  Technical Success | 894 | 138
  Procedural Success | 892 | 138

7. Secondary Outcome: Number of Participants With Freedom From Target Lesion Revascularization (TLR) at 6, 12, and 24 Months Post Index Procedure
Time Frame: 6, 12, and 24 months post index procedure
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lutonix Drug Coated Balloon | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 981 | 153
participants
  6 months post index procedure | 940 | 144
  12 months post index procedure: number analyzed (Participants) | 955 | 146
  12 months post index procedure | 839 | 122
  24-Months Post-Index Procedure: number analyzed (Participants) | 898 | 138
  24-Months Post-Index Procedure | 706 | 104

8. Secondary Outcome: Number of Participants With Alternative Primary Patency at 6, 12, and 24 Months Post Index Procedure
Description: Percentage of subjects with Alternative Primary Patency based on alternative definitions of duplex ultrasound (DUS) peak systolic velocity ratio (PSVR) <2.0 and <3.0 at 6, 12, and 24 months post index procedure. DUS PSVR was calculated by dividing the maximum peak systolic velocity (PSV) from the stenosis by the PSV from the nearest segment of normal artery above the site of increase.
Time Frame: 6, 12, and 24 months post index procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix Drug Coated Balloon | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 792 | 136
Participants
  DUS PSVR >=2.0: 6 months post index procedure: number analyzed (Participants) | 790 | 135
  DUS PSVR >=2.0: 6 months post index procedure | 565 | 74
  DUS PSVR >=2.0: 12 months post index procedure: number analyzed (Participants) | 762 | 133
  DUS PSVR >=2.0: 12 months post index procedure | 400 | 62
  DUS PSVR >=2.0: 24 months post index procedure: number analyzed (Participants) | 716 | 113
  DUS PSVR >=2.0: 24 months post index procedure | 282 | 38
  DUS PSVR >=3.0: 6 months post index procedure | 670 | 98
  DUS PSVR >=3.0: 12 months post index procedure: number analyzed (Participants) | 743 | 127
  DUS PSVR >=3.0: 12 months post index procedure | 492 | 73
  DUS PSVR >=3.0: 24 months post index procedure: number analyzed (Participants) | 671 | 105
  DUS PSVR >=3.0: 24 months post index procedure | 344 | 48

9. Secondary Outcome: Improvement in Rutherford Classification Scores at 6, 12, and 24 Months Post Index Procedure Compared to Baseline
Description: The endpoint summarizes the change in index-limb Rutherford Classification of participants from baseline through 24 months. Data is presented as shift from baseline Rutherford Classification data using the following categories: 1) Improvement, 2) Same, and 3) Worsened.
Time Frame: 6, 12, and 24 months post index procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix Drug Coated Balloon | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 944 | 145
Participants
  6 months from baseline: Improved | 830 | 118
  6 months from baseline: Same | 79 | 22
  6 months from baseline: Worsened | 35 | 5
  12 months from baseline: number analyzed (Participants) | 890 | 131
  12 months from baseline: Improved | 771 | 108
  12 months from baseline: Same | 89 | 21
  12 months from baseline: Worsened | 30 | 2
  24 months from baseline: number analyzed (Participants) | 816 | 122
  24 months from baseline: Improved | 701 | 106
  24 months from baseline: Same | 88 | 15
  24 months from baseline: Worsened | 27 | 1

10. Secondary Outcome: Change in Resting Ankle Brachial Index (ABI) at 6, 12, and 24 Months Compared to Baseline
Description: Mean change from baseline values. The Ankle Brachial Index (ABI) is defined as a ratio of ankle to brachial (upper arm) artery systolic blood pressure and aims at determining how well the blood is flowing in the legs.
Time Frame: 6, 12, and 24 months from baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Lutonix Drug Coated Balloon | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 892 | 135
Ratio
  6 months post index procedure | 0.19 (0.26) | 0.16 (0.22)
  12 months post index procedure: number analyzed (Participants) | 845 | 126
  12 months post index procedure | 0.18 (0.26) | 0.18 (0.25)
  24-Months Post-Index Procedure: number analyzed (Participants) | 753 | 112
  24-Months Post-Index Procedure | 0.16 (0.27) | 0.17 (0.24)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and Serious Adverse Events (SAEs) collected by all sites from the time of index procedure to 60 months follow up.
Arm/Group | Lutonix Drug Coated Balloon | Standard Uncoated Angioplasty Balloon
All-Cause Mortality (participants affected / at risk) | 147/1029 | 17/160
Serious Adverse Events (participants affected / at risk) | 813/1029 | 125/160
Other Adverse Events (participants affected / at risk) | 845/1029 | 126/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lutonix Drug Coated Balloon (N=1029) | Standard Uncoated Angioplasty Balloon (N=160)
Arterial occlusion puncture site (General disorders) | 1 | 0
Hematoma / bleeding puncture site - major (General disorders) | 8 | 1
Hematoma / bleeding puncture site - minor (General disorders) | 8 | 0
Pseudo aneurysm (General disorders) | 9 | 2
Puncture site infection (General disorders) | 2 | 0
Vascular perforation / rupture (General disorders) | 1 | 0
Retroperitoneal bleed (General disorders) | 3 | 1
Significant blood loss (General disorders) | 1 | 0
Other Access site complication (General disorders) | 7 | 0 — This category of SAEs is not broken down further in the Clinical Study Report.
Acute coronary syndrome (Vascular disorders) | 23 | 2 — Category "Cardiovascular" in Clinical Study Report.
Angina, stable (Vascular disorders) | 65 | 8 — Category "Cardiovascular" in Clinical Study Report.
Angina, unstable (Vascular disorders) | 58 | 5 — Category "Cardiovascular" in Clinical Study Report.
Arrhythmia - Bradycardia (Vascular disorders) | 22 | 3 — Category "Cardiovascular" in Clinical Study Report.
Arrhythmia - Tachycardia (Vascular disorders) | 20 | 6 — Category "Cardiovascular" in Clinical Study Report.
Arrhythmia - Other (Vascular disorders) | 45 | 10 — Category "Cardiovascular" in Clinical Study Report. This category is not broken down further in the Clinical Study Report.
Cardiac tamponade (Vascular disorders) | 1 | 0 — Category "Cardiovascular" in Clinical Study Report.
Cardiogenic shock (Vascular disorders) | 9 | 1 — Category "Cardiovascular" in Clinical Study Report.
Chronic heart failure (Vascular disorders) | 59 | 8 — Category "Cardiovascular" in Clinical Study Report.
Death (Vascular disorders) | 17 | 1 — Category "Cardiovascular" in Clinical Study Report.
Endocarditis (Vascular disorders) | 2 | 0 — Category "Cardiovascular" in Clinical Study Report.
Hypertension (Vascular disorders) | 33 | 10 — Category "Cardiovascular" in Clinical Study Report.
Hypotension (Vascular disorders) | 14 | 0 — Category "Cardiovascular" in Clinical Study Report.
Myocardial infarction (Vascular disorders) | 69 | 17 — Category "Cardiovascular" in Clinical Study Report.
Other Cardiovascular (Vascular disorders) | 152 | 20 — Category "Cardiovascular" in Clinical Study Report.
Diabetes Mellitus, Type I (Endocrine disorders) | 3 | 0
Diabetes Mellitus, Type II (Endocrine disorders) | 12 | 2
Hyperthroidism (Endocrine disorders) | 1 | 0
Hypothroidism (Endocrine disorders) | 1 | 0
Other Endocrine system (Endocrine disorders) | 16 | 2 — These SAEs are not broken down further in the Clinical Study Report.
Cholecystitis (Gastrointestinal disorders) | 17 | 4
Colon carcinoma (Gastrointestinal disorders) | 3 | 2
Diarrhea (Gastrointestinal disorders) | 15 | 6
Epigastric pain (Gastrointestinal disorders) | 3 | 3
Gastritis (Gastrointestinal disorders) | 8 | 1
Gastrointestinal bleeding (Gastrointestinal disorders) | 46 | 8
Nausea (Gastrointestinal disorders) | 4 | 1
Other infections / inflammatory (Gastrointestinal disorders) | 11 | 0 — Category of SAE not otherwise broken down in the Clinical Study Report.
Other infectious / inflammatory (Gastrointestinal disorders) | 3 | 2 — Category of SAE not otherwise broken down in the Clinical Study Report.
Pancreatitis (Gastrointestinal disorders) | 11 | 3
Peritonitis (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 8 | 2
Other Gastrointestinal (Gastrointestinal disorders) | 68 | 11 — Category of SAE not otherwise broken down in the Clinical Study Report.
Local infection (Infections and infestations) | 30 | 8
Septic shock (Infections and infestations) | 1 | 0
Septicemia / bacteremia (Infections and infestations) | 18 | 1
Other Infectious (Infections and infestations) | 23 | 3 — Category of SAE not otherwise broken down in the Clinical Study report.
Confusion (Nervous system disorders) | 8 | 3 — Category "Neurological/Nervous System" in Clinical Study Report.
Death (Nervous system disorders) | 1 | 0 — Category "Neurological/Nervous System" in Clinical Study Report.
Depression (Nervous system disorders) | 6 | 1 — Category "Neurological/Nervous System" in Clinical Study Report.
Dizziness / vertigo (Nervous system disorders) | 8 | 1 — Category "Neurological/Nervous System" in Clinical Study Report.
Fainting / syncope (Nervous system disorders) | 17 | 3 — Category "Neurological/Nervous System" in Clinical Study Report.
Peripheral nervous system complication (Nervous system disorders) | 4 | 1 — Category "Neurological/Nervous System" in Clinical Study Report.
Seizure (Nervous system disorders) | 4 | 1 — Category "Neurological/Nervous System" in Clinical Study Report.
Stroke - hemorrhagic (Nervous system disorders) | 6 | 1 — Category "Neurological/Nervous System" in Clinical Study Report.
Stroke - ischemic (Nervous system disorders) | 36 | 3 — Category "Neurological/Nervous System" in Clinical Study Report.
TIA (Nervous system disorders) | 26 | 2 — Category "Neurological/Nervous System" in Clinical Study Report.
Other Neurological / nervous system (Nervous system disorders) | 43 | 7 — Category of SAE not otherwise broken down in the Clinical Study Report. Category "Neurological/Nervous System" in Clinical Study Report.
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 15 | 2
Carcinoma (Respiratory, thoracic and mediastinal disorders) | 27 | 3
COPD (Respiratory, thoracic and mediastinal disorders) | 39 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Death (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Other respiratory (Respiratory, thoracic and mediastinal disorders) | 43 | 6 — Category of SAE not otherwise broken down in Clinical Study Report.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 75 | 7
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 0 — Category "Skeletal, Spine and Muscular System" in Clinical Study Report.
Arthritis (Musculoskeletal and connective tissue disorders) | 13 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 4
Fracture (bone) (Musculoskeletal and connective tissue disorders) | 47 | 10
Hernia (Musculoskeletal and connective tissue disorders) | 20 | 0
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 12 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Claudication (Musculoskeletal and connective tissue disorders) | 12 | 6
Other Skeletal, spine and muscular system (Musculoskeletal and connective tissue disorders) | 89 | 12 — Category of SAE not otherwise broken down in Clinical Study report.
Allergy (General disorders) | 1 | 0 — SAE entered as part of a Category titled "Systematic Complication" in Clinical Study Report.
Anaphylatic reaction (General disorders) | 3 | 1 — SAE entered as part of a Category titled "Systematic Complication" in Clinical Study Report.
Other Systematic complication (General disorders) | 6 | 0 — Category of SAE not further broken down in Clinical Study Report. SAE entered as part of a Category titled "Systematic Complication" in Clinical Study Report.
Aneurysm (General disorders) | 1 | 0 — This SAE was entered in "Target Vessel" category in Clinical Study Report.
Atherosclerosis (General disorders) | 15 | 4 — This SAE was entered in "Target Vessel" category in Clinical Study Report.
Dissection (General disorders) | 3 | 0 — This SAE was entered in "Target Vessel" category in Clinical Study Report.
Embolism (General disorders) | 1 | 0 — This SAE was entered in "Target Vessel" category in Clinical Study Report.
Occlusion / closure (General disorders) | 18 | 5 — This SAE was entered in "Target Vessel" category in Clinical Study Report.
Perforation (General disorders) | 2 | 0 — This SAE was entered in "Target Vessel" category in Clinical Study Report.
Restenosis (General disorders) | 65 | 18 — This SAE was entered in "Target Vessel" category in Clinical Study Report.
Thrombus - in-lesion (General disorders) | 1 | 2 — This SAE was entered in "Target Vessel" category in Clinical Study Report.
Other Target vessel (General disorders) | 10 | 1 — This SAE was entered in "Target Vessel" category in Clinical Study Report. SAE not otherwise broken down in the Clinical Study Report.
Bladder infection (Renal and urinary disorders) | 4 | 0 — SAE part of a category titled "Genito-urinary" in Clinical Study report.
Kidney stones (Renal and urinary disorders) | 5 | 0 — SAE part of a category titled "Genito-urinary" in Clinical Study report.
Prostate carcinoma (Renal and urinary disorders) | 5 | 1 — SAE part of a category titled "Genito-urinary" in Clinical Study report.
Prostate hypertrophy (Renal and urinary disorders) | 7 | 0 — SAE part of a category titled "Genito-urinary" in Clinical Study report.
Renal failure / insufficiency (Renal and urinary disorders) | 54 | 9 — SAE part of a category titled "Genito-urinary" in Clinical Study report.
Urinary infection (Renal and urinary disorders) | 21 | 5 — SAE part of a category titled "Genito-urinary" in Clinical Study report.
Urinary retention (Renal and urinary disorders) | 2 | 1 — SAE part of a category titled "Genito-urinary" in Clinical Study report.
Other Genito-urinary system (Renal and urinary disorders) | 48 | 5 — SAE part of a category titled "Genito-urinary" in Clinical Study report. SAE entry not otherwise broken down in Clinical Study Report.
Abscess (General disorders) | 6 | 0 — SAE entered in a category titled "Various" in the Clinical Study Report. Therefore, the SAE is hereby classified under "General Disorder" Organ System category.
Amputation (General disorders) | 8 | 1 — SAE entered in a category titled "Various" in the Clinical Study Report. Therefore, the SAE is hereby classified under "General Disorder" Organ System category.
Atypical chest pain (General disorders) | 7 | 2 — SAE entered in a category titled "Various" in the Clinical Study Report. Therefore, the SAE is hereby classified under "General Disorder" Organ System category.
Carcinoma (not specified elsewhere) (General disorders) | 58 | 5 — SAE entered in a category titled "Various" in the Clinical Study Report. Therefore, the SAE is hereby classified under "General Disorder" Organ System category.
Death (non-cardiac or neurological) (General disorders) | 23 | 1 — SAE entered in a category titled "Various" in the Clinical Study Report. Therefore, the SAE is hereby classified under "General Disorder" Organ System category.
Fatigue (General disorders) | 2 | 2 — SAE entered in a category titled "Various" in the Clinical Study Report. Therefore, the SAE is hereby classified under "General Disorder" Organ System category.
Fever (General disorders) | 4 | 0 — SAE entered in a category titled "Various" in the Clinical Study Report. Therefore, the SAE is hereby classified under "General Disorder" Organ System category.
Headache (General disorders) | 1 | 0 — SAE entered in a category titled "Various" in the Clinical Study Report. Therefore, the SAE is hereby classified under "General Disorder" Organ System category.
Hematuria (General disorders) | 3 | 0 — SAE entered in a category titled "Various" in the Clinical Study Report. Therefore, the SAE is hereby classified under "General Disorder" Organ System category.
Rash (General disorders) | 1 | 0 — SAE entered in a category titled "Various" in the Clinical Study Report. Therefore, the SAE is hereby classified under "General Disorder" Organ System category.
Sepsis (General disorders) | 7 | 1 — SAE entered in a category titled "Various" in the Clinical Study Report. Therefore, the SAE is hereby classified under "General Disorder" Organ System category.
Other (General disorders) | 163 | 21 — SAE entered in a category titled "Various" in the Clinical Study Report. Therefore, the SAE is hereby classified under "General Disorder" Organ System category. SAE "other" is not otherwise broken down in the Clinical Study Report.
Aneurysm (General disorders) | 7 | 1 — SAE entered in category "Vessel specific complications in the leg (not target lesion or target vessel)" in Clinical Study Report.
Arterial occlusion (General disorders) | 36 | 9 — SAE entered in category "Vessel specific complications in the leg (not target lesion or target vessel)" in Clinical Study Report.
Arterial thrombosis (General disorders) | 6 | 2 — SAE entered in category "Vessel specific complications in the leg (not target lesion or target vessel)" in Clinical Study Report.
Atherosclerosis (General disorders) | 36 | 11 — SAE entered in category "Vessel specific complications in the leg (not target lesion or target vessel)" in Clinical Study Report.
Dissection (General disorders) | 3 | 0 — SAE entered in category "Vessel specific complications in the leg (not target lesion or target vessel)" in Clinical Study Report.
Embolism (General disorders) | 7 | 0 — SAE entered in category "Vessel specific complications in the leg (not target lesion or target vessel)" in Clinical Study Report.
Hematoma / bleeding (General disorders) | 2 | 0 — SAE entered in category "Vessel specific complications in the leg (not target lesion or target vessel)" in Clinical Study Report.
Perforation (General disorders) | 1 | 0 — SAE entered in category "Vessel specific complications in the leg (not target lesion or target vessel)" in Clinical Study Report.
Restenosis (General disorders) | 112 | 22 — SAE entered in category "Vessel specific complications in the leg (not target lesion or target vessel)" in Clinical Study Report.
Stent thrombosis (definite) (General disorders) | 4 | 2 — SAE entered in category "Vessel specific complications in the leg (not target lesion or target vessel)" in Clinical Study Report.
Stent thrombosis (possible) (General disorders) | 2 | 1 — SAE entered in category "Vessel specific complications in the leg (not target lesion or target vessel)" in Clinical Study Report.
Venous occlusion (General disorders) | 2 | 0 — SAE entered in category "Vessel specific complications in the leg (not target lesion or target vessel)" in Clinical Study Report.
Venous thrombosis (General disorders) | 7 | 2 — SAE entered in category "Vessel specific complications in the leg (not target lesion or target vessel)" in Clinical Study Report.
Ischemia (General disorders) | 5 | 2 — SAE entered in category "Vessel specific complications in the leg (not target lesion or target vessel)" in Clinical Study Report.
Stenosis (General disorders) | 126 | 23 — SAE entered in category "Vessel specific complications in the leg (not target lesion or target vessel)" in Clinical Study Report.
Other Vessel Specific (General disorders) | 22 | 2 — SAE entered in category "Vessel specific complications in the leg (not target lesion or target vessel)" in Clinical Study Report. SAE not otherwise broken down in the Clinical Study report.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lutonix Drug Coated Balloon (N=1029) | Standard Uncoated Angioplasty Balloon (N=160)
Hematoma / bleeding puncture site - minor (General disorders) | 51 | 4 — AE entered in category "Access Site Complication" in the Clinical Study Report.
Angina, Stable (Cardiac disorders) | 46 | 11 — AE entered in category "Cardiovascular" in clinical Study report.
Arrhythmia - Other (Cardiac disorders) | 47 | 10 — AE entered in category "Cardiovascular" in clinical Study report. AE (other) not otherwise broken down in Clinical Study Report.
Hypertension (Cardiac disorders) | 64 | 9 — AE entered in category "Cardiovascular" in clinical Study report.
Hypotension (Cardiac disorders) | 32 | 3 — AE entered in category "Cardiovascular" in clinical Study report.
Other Cardiovascular (Cardiac disorders) | 110 | 23 — AE entered in category "Cardiovascular" in clinical Study report. AE "Other" not otherwise broken down in the Clinical Study report.
Diabetes Mellitus, Type II (Endocrine disorders) | 35 | 7
Other Endocrine system (Endocrine disorders) | 33 | 3 — AE (Other) not otherwise broken down in Clinical Study Report.
Nausea (Gastrointestinal disorders) | 31 | 2
Other Gastrointestinal (Gastrointestinal disorders) | 118 | 11 — AE (other) not otherwise broken down in Clinical Study Report.
Local infection (Infections and infestations) | 72 | 12
Other infectious (Infections and infestations) | 43 | 4 — AE (Other) not otherwise broken down in the Clinical Study Report.
Dizziness / vertigo (Nervous system disorders) | 46 | 9
Other Neurological / nervous system (Nervous system disorders) | 92 | 13 — AE (Other) not otherwise broken down in the Clinical Study Report.
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 46 | 5
COPD (Respiratory, thoracic and mediastinal disorders) | 31 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 44 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 53 | 7
Other respiratory (Respiratory, thoracic and mediastinal disorders) | 88 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 43 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 38 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 112 | 8
Fracture (bone) (Musculoskeletal and connective tissue disorders) | 42 | 7
Claudication (Musculoskeletal and connective tissue disorders) | 79 | 17
Other skeletal, spine and muscular system (Musculoskeletal and connective tissue disorders) | 272 | 35 — AE (Other) not otherwise broken down in Clinical Study Report.
Dissection (General disorders) | 26 | 6 — AE entered in "Target Lesion" Category of Clinical Study Report.
Restenosis (General disorders) | 53 | 11
Renal failure / insufficiency (Renal and urinary disorders) | 57 | 5
Urinary infection (Renal and urinary disorders) | 72 | 9
Other Genito-urinary system (General disorders) | 52 | 13 — AE (Other) not otherwise broken down in the Clinical Study Report.
Rash (General disorders) | 41 | 5 — AE reported in category "Various" in the Clinical Study Report.
Other (General disorders) | 399 | 67 — AE "Other" not otherwise broken down in the Clinical Study Report.
Restenosis (General disorders) | 31 | 3 — AE reported in category "Vessel specific complications in the leg (not target lesion or target vessel)"in the Clinical Study Report.
Stenosis (General disorders) | 40 | 5 — AE reported in category "Vessel specific complications in the leg (not target lesion or target vessel)"in the Clinical Study Report.
Other Vessel Specific (General disorders) | 55 | 13 — AE reported in category "Vessel specific complications in the leg (not target lesion or target vessel)"in the Clinical Study Report. AE (Other) not otherwise broken down in clinical Study Report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-12-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT01790243/Prot_SAP_000.pdf